CLINICAL TRIAL: NCT06161714
Title: The Effectiveness of Buccal Infiltration Only Using Articaine for Routine Exodontia of Mandibular Molar: A Cross-Over Randomized Controlled Clinical Trial
Brief Title: The Effectiveness of Buccal Infiltration Only Using Articaine for Extraction of Mandibular Molar
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Albatool Baroom, Resident of Oral & Maxillofacial Surgery in postgraduate program in Riyadh El University, Riyadh Elm University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FPGRP/2023/791/1041
Record Dates: First submitted 2023-11-25; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Carticaine; Epinephrine; Lidocaine

STUDY DESIGN:
Intervention Model Description: One 1.8 ml cartridge of 4% articaine with 1:100,000 epinephrine will be utilized in the articaine group and one 1.8 ml cartridge of 2% lidocaine with 1:100,000 epinephrine will be utilized in the lidocaine group. The cartridges will be of similar size and shape, to be allotted a special code, enclosed in thin, adhesive tape by the distributor, and kept into one box for articaine and another box for lidocaine.
  A 27-gauge needle will be used for buccal infiltration in each case. Any sensation of pain after administering the local anesthesia will be considered as a failure and an inferior alveolar nerve block will be given. Otherwise, the tooth will be extracted with no additional anesthesia.
Who Masked: Participant, Investigator
Masking Description: This is a double blinded randomized clinical trial, which neither the injector (investigator) nor the participant will know what anesthesia type was used in each session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Right mandibular molar (Experimental): Articaine 4% with 1:100,000 epinephrine
  Interventions: Drug: Articaine 4%/Epi 1:100000 Inj Cart 1.7Ml
- Left mandibular molar (Experimental): Lidocaine 2% with 1:100,000
  Interventions: Drug: Lidocaine 2%/Epi 1:100000 Inj Cart 1.7Ml

INTERVENTIONS:
Drug: Articaine 4%/Epi 1:100000 Inj Cart 1.7Ml — 4% articaine with 1:100,000 epinephrine buccal infiltration
  Other Names: Septanest
  Arms: Right mandibular molar
Drug: Lidocaine 2%/Epi 1:100000 Inj Cart 1.7Ml — 2% Lidocaine with 1:100,000 epinephrine buccal infiltration
  Other Names: Octocaine
  Arms: Left mandibular molar

SUMMARY:
The goal of this clinical trial, is to test out the efficacy of using Articaine only as a local anesthesia as buccal infiltration to extract lower molar teeth.

Study will be performed in patients visiting Riyadh Elm University clinics seeking extraction of lower molars bilaterally, in each visit one molar tooth will be extracted using Ariticaine and the second visit with Lidocaine, pain level will be monitored and documented.

This study may be helpful in providing scientific information to the oral maxillofacial surgeons which will assist them in choosing the best local anesthetic agent, and possibly substituting using inferior alveolar nerve block with infiltration only when extracting the mandibular posterior teeth.

DETAILED DESCRIPTION:
This is a double-blind, randomized clinical trial, which will involve 40 patients visiting the out-patient department of Oral and Maxillofacial surgery. For each patient, one mandibular molar will be extracted from right as well as left side, with one side being anesthetized using 4% articaine with 1:100,000 epinephrine and other with 2% lidocaine with 1:100,000 epinephrine buccal infiltration only. Evaluation and comparison will be done on the basis of pain prevalence exhibited by the patients while extraction.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Patients with age more than 18 years
* Patients indicated for at least one mandibular molar extraction
* Patients with the ability to fill the questionnaire

Exclusion Criteria:

* Patients with abscess or any lesion, which may affect the local anesthesia provision.
* Patients with stage III mobile teeth
* Patients with a history of medical conditions such as diabetes mellitus, heart disease, pregnancy, allergy or renal disease
* Patients who are not able to give an informed consent or are not agreeing to take part in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-04-10 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain measurement | Pain will be measured after injection, during extraction procedure and at the end of the session immediately after finishing the procedure, scale of pain will be 0 for no pain and 10 for maximum pain
  Pain will be measured using the vial analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Albatool Baroom, Principal Investigator — Albatool.a.baroom2021@student.riyadh.edu.sa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Averbuch M, Katzper M. Assessment of visual analog versus categorical scale for measurement of osteoarthritis pain. J Clin Pharmacol. 2004 Apr;44(4):368-72. doi: 10.1177/0091270004263995. PMID 15051743
- [Result] Bartlett G, Mansoor J. Articaine buccal infiltration vs lidocaine inferior dental block - a review of the literature. Br Dent J. 2016 Feb 12;220(3):117-20. doi: 10.1038/sj.bdj.2016.93. PMID 26868800
- [Result] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Result] Kanaa MD, Whitworth JM, Corbett IP, Meechan JG. Articaine and lidocaine mandibular buccal infiltration anesthesia: a prospective randomized double-blind cross-over study. J Endod. 2006 Apr;32(4):296-8. doi: 10.1016/j.joen.2005.09.016. Epub 2006 Feb 17. PMID 16554198
- [Result] Majid OW, Muhammad ZA. Effectiveness of Articaine Buccal Infiltration Anesthesia for Mandibular Premolar Extraction: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. J Oral Maxillofac Surg. 2019 Sep;77(9):1784-1789. doi: 10.1016/j.joms.2019.03.033. Epub 2019 Mar 30. PMID 31028737
- [Result] Myles PS, Myles DB, Galagher W, Boyd D, Chew C, MacDonald N, Dennis A. Measuring acute postoperative pain using the visual analog scale: the minimal clinically important difference and patient acceptable symptom state. Br J Anaesth. 2017 Mar 1;118(3):424-429. doi: 10.1093/bja/aew466. PMID 28186223
- [Result] Rathi NV, Khatri AA, Agrawal AG, M SB, Thosar NR, Deolia SG. Anesthetic Efficacy of Buccal Infiltration Articaine versus Lidocaine for Extraction of Primary Molar Teeth. Anesth Prog. 2019 Spring;66(1):3-7. doi: 10.2344/anpr-65-04-02. PMID 30883236
- [Result] Rayati F, Noruziha A, Jabbarian R. Efficacy of buccal infiltration anaesthesia with articaine for extraction of mandibular molars: a clinical trial. Br J Oral Maxillofac Surg. 2018 Sep;56(7):607-610. doi: 10.1016/j.bjoms.2018.06.012. Epub 2018 Jul 3. PMID 29980352
- [Result] Robertson D, Nusstein J, Reader A, Beck M, McCartney M. The anesthetic efficacy of articaine in buccal infiltration of mandibular posterior teeth. J Am Dent Assoc. 2007 Aug;138(8):1104-12. doi: 10.14219/jada.archive.2007.0324. PMID 17670879
- [Result] Soysa NS, Soysa IB, Alles N. Efficacy of articaine vs lignocaine in maxillary and mandibular infiltration and block anesthesia in the dental treatments of adults: A systematic review and meta-analysis. J Investig Clin Dent. 2019 Aug;10(3):e12404. doi: 10.1111/jicd.12404. Epub 2019 Mar 18. PMID 30887677
- [Result] Thiem DGE, Schnaith F, Van Aken CME, Kontges A, Kumar VV, Al-Nawas B, Kammerer PW. Extraction of mandibular premolars and molars: comparison between local infiltration via pressure syringe and inferior alveolar nerve block anesthesia. Clin Oral Investig. 2018 Apr;22(3):1523-1530. doi: 10.1007/s00784-017-2251-7. Epub 2017 Oct 17. PMID 29043507